CLINICAL TRIAL: NCT06183580
Title: Neurofeedback and Neural Plasticity of Self-Processing and Affect Regulation Circuits in Suicide Attempting Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSYCH-2020-29400
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Suicide, Attempted; Suicide, Ideation; Depression
MeSH Terms: conditions — Suicide, Attempted; Suicide; Depression

STUDY DESIGN:
Intervention Model Description: Comparing two different targets of treatment: either amygdala or dorsal anterior cingulate cortex neurofeedback
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dACC Arm (Experimental): Participants assigned to the Neurofeedback from the dorsal anterior cingulate cortex
  Interventions: Other: neurofeedback training involving dACC
- rAMY Arm (Experimental): Participants assigned to the Neurofeedback from the amygdala
  Interventions: Other: neurofeedback training involving amygdala

INTERVENTIONS:
Other: neurofeedback training involving dACC — Participants are pseudorandomized to the dACC group to undergo neurofeedback (NF). NF training consists of four ~7.33 min NF training runs preceded by a 5 min baseline (no NF) and followed by a 5 min transfer run (no NF). Training entails NF blocks paired to a self-happy face along a bar that indicates changing levels of the dACC. During the control condition, participants will count backward (CB) from 100 cued by an unfamiliar happy face with no NF. During rest conditions, participants see the cue "Rest" and are asked to relax with their eyes open. During NF, participants will try to increase dACC neural activity by recalling happy memories. The colored bar indicating the neural activity will shift up or down depending on values provided by Turbo-BrainVoyager software. Green = Activity > baseline and red = Activity < baseline. Before and after NF training, suicide ideation severity, depression severity, and performance on self-processing behavioral tasks will be assessed.
  Arms: dACC Arm
Other: neurofeedback training involving amygdala — Participants are pseudorandomized to the rAMY group to undergo neurofeedback (NF). NF training consists of four ~7.33 min NF training runs preceded by a 5 min baseline (no NF) and followed by a 5 min transfer run (no NF). Training entails NF blocks paired to a self-happy face along a bar that indicates changing levels of the rAMY. During the control condition, participants will count backward (CB) from 100 cued by an unfamiliar happy face with no NF. During rest conditions, participants see the cue "Rest" and are asked to relax with their eyes open. During NF, participants will try to increase rAMY neural activity by recalling happy memories. The colored bar indicating the neural activity will shift up or down depending on values provided by Turbo-BrainVoyager software. Green = Activity > baseline and red = Activity < baseline. Before and after NF training, suicide ideation severity, depression severity, and performance on self-processing behavioral tasks will be assessed.
  Arms: rAMY Arm

SUMMARY:
A non invasive treatment study including participants at risk for suicide attempts and undergoing neurofeedback training. Neurofeedback is controlling your brain activity in real time inside the scanner.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with a history of suicide attempts

Exclusion Criteria:

* Psychotic disorders.
* Primary substance use disorder.
* Primary anorexic disorder.
* Autism Spectrum Disorder.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-28 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
suicide ideation | 1 week and 1 month following intervention
  suicide ideation questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Karina Quevedo, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT06183580/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT06183580/ICF_001.pdf